CLINICAL TRIAL: NCT01636505
Title: The Results of Preimplantation Genetic Diagnosis and Preimplantation Genetic Screening of Embryos Obtained From GnRH-agonist Long and GnRH-antagonist Ovarian Stimulation Protocol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ECK011170
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Embryo's Genetic and Chromosomal Quality
MeSH Terms: interventions — cetrorelix; ganirelix; Gonadotropin-Releasing Hormone; Buserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- short protocol (Active Comparator): gnrh agonist versus gnrh antagonist
  Interventions: Drug: ghrh antagonist (cetrotide/orgalutran)
- long protocol (Active Comparator)
  Interventions: Drug: gnrh agonist (suprefact)

INTERVENTIONS:
Drug: ghrh antagonist (cetrotide/orgalutran) — cetrotide/orgalutran 0.25 mg
  Arms: short protocol
Drug: gnrh agonist (suprefact) — suprefact 5.5 ml
  Arms: long protocol

SUMMARY:
The aim of this study is to performed a randomized controlled trial to evaluate the rate of genetic and chromosomal abnormalities in embryos obtained from GnRH-agonist long and GnRH-antagonist ovarian stimulation protocols.

Patients will be prospectively randomized in two groups: the first undergoing controlled ovarian stimulation in GnRH-agonist long protocol and the second following GnRH-antagonist ovarian stimulation regimen.

The end-points of the study include the number of genetically and chromosomally abnormal embryos, the pregnancy, the implantation and the healthy baby birth rate.

The patients included in PGS program were selected on the base of advanced maternal age, repeated pregnancy lost and implantation failure whereas the patients who were know to carry sex-linked or monogenic disorders were considered for PGD strategy.

The uterine abnormalities, endometriosis and endocrinal diseases were considered to be the exclusion factors.

ELIGIBILITY:
Inclusion Criteria:

* patients carrier genetic disease
* advanced maternal Age
* repeated IVF failure
* recurrent pregnancy loss

Exclusion Criteria:

* uterine abnormalities
* endometriosis
* endocrinal diseases

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The results of Preimplantation Genetic Diagnosis and Preimplantation Genetic Screening of embryos obtained from GnRH-agonist long and GnRH-antagonist ovarian stimulation protocol | one year
  difference in embryos' genetic and chromosomal quality using two different ovarian stimulation protocol

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy